CLINICAL TRIAL: NCT00916578
Title: A Phase II Study of Preoperative Capecitabine and Concomitant Radiation in Women With Advanced Inflammatory or Non-Inflammatory Breast Cancer
Brief Title: Xeloda (Capecitabine) and External Beam Radiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0087; NCI-2012-01266 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Advanced Inflammatory Breast Cancer; Non-Inflammatory Breast Cancer; Capecitabine; Xeloda; Concomitant Radiation; Radiation Therapy; Radiotherapy; Women
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy + Capecitabine (Experimental): Capecitabine 825 mg/m2 twice a day. One of the two daily doses of capecitabine should be taken approximately 2 hours before receiving radiotherapy. The first day of Capecitabine is same day that radiotherapy is started, and last day that Capecitabine is given is last day of radiotherapy. Capecitabine administered only on days patient receives radiation therapy.
  Radiation therapy dose 50-57 Gy to initial clinical target volume (CTV, gross disease + tissue at risk for micrometastatic disease including margin around gross disease and draining regional lymphatics).
  Interventions: Radiation: Radiation Therapy; Drug: Capecitabine

INTERVENTIONS:
Radiation: Radiation Therapy — 50-57 Gy per faction once or twice a day, 5 days a week, for about 5 -7 weeks, about 15-30 minutes each time.
  Other Names: RT; Radiotherapy
Drug: Capecitabine — During 5-7 weeks of radiation therapy, 825 mg/m2 (pills) by mouth, 2 times a day, about 12 hours apart, 30 minutes after eating food and about 2 hours before radiation therapy.
  Other Names: Xeloda

SUMMARY:
The goal of this clinical research study is to find out if Xeloda® (capecitabine) and radiation therapy can help to control breast cancer that did not respond well to chemotherapy.

The safety of this study treatment will also be studied.

DETAILED DESCRIPTION:
The Study Treatment:

Radiation therapy and capecitabine are both designed to interfere with the growth of cancer cells.

Study Therapy:

If you are found to be eligible to take part in this study, you will receive radiation therapy once or twice a day, 5 days a week, for about 5 -7 weeks. The schedule and number of weeks will be the doctor's decision based on the type of breast cancer.

The radiation treatments will take about 15-30 minutes each time.

You will take the Capecitabine pills by mouth every day during the 5-7 weeks that you receive radiation therapy. The pills should be taken 2 times a day, about 12 hours apart, 30 minutes after eating food. On the radiation therapy days, you will take capecitabine about 2 hours before the radiation therapy.

You will be given a pill diary in which you should record what time you take each dose of capecitabine.

Study Visits:

Once a week while you are receiving study treatment, you will have a physical exam.

Length of Study:

You may remain on study treatment for up to 7 weeks. You will be taken off study treatment early if the disease gets worse or intolerable side effects occur.

Based on the status of the cancer, if you become eligible to have surgery after radiation, you will be referred to a surgeon to discuss that option.

Follow-Up Visits:

At Month 3 after finishing radiation therapy (or surgery, if applicable), you will have a positron emission tomography / computed tomography (PET/CT) scan or ultrasound to check the status of the disease.

At Months 9, 17, and 29 after finishing radiation therapy or surgery, you may have a PET/CT scan, ultrasound, and/or routine blood tests if your doctor thinks it is needed. The amount of blood drawn, if any, will be the doctor's decision based on routine care.

This is an investigational study. Capecitabine is commercially available and FDA approved to treat breast cancer that has spread. Radiation therapy is also commonly used to treat breast cancer. The combination of capecitabine and radiation therapy is commonly used to treat rectal cancer.

At this time, it is considered investigational to give the combination of capecitabine and radiation therapy to patients with breast cancer.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of invasive breast cancer
2. No contraindications to receiving a course of radiation treatment (pregnancy, prior radiation to the volume with disease, or systemic disease in which radiation therapy is an absolute contraindication)
3. Patients who have chemo-refractory gross disease in the breast causing symptoms (pain, drainage, duress) OR gross disease in the breast (greater than or equal to T3) and/or lymph node(s) progressive, persistent, or minimally responsive to chemotherapy deemed inoperable or questionable inoperable OR Recurrent gross disease in a previously unirradiated breast or on the chest wall or in the regional lymphatics (core biopsy will not be offered to patients without gross disease in the breast).
4. Are able to swallow and retain oral medication (intact pill)
5. Age over 18
6. Female gender

Exclusion Criteria:

1. Have an active or uncontrolled infection
2. Have dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
3. Have used an investigational drug within 21 days preceding the first dose of study medication
4. Are receiving therapeutic anti-coagulation therapy (i.e. warfarin, heparin)
5. Uncontrolled arrhythmia or congestive heart failure (CHF) based on clinical history or physical exam
6. Patient cannot receive whole brain irradiation concurrently with Xeloda treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-06-05 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Woodward, MD, PHD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary objective is to determine the rate of responses by RECIST criteria in all patients who received treatment that includes pre-operative or palliative concurrent radiation with capecitabine to the breast and at risk or involved regional lymph node basins. The recruitment process was located at MD Anderson Cancer Center between 2009 to 2012.
Groups:
- Single Arm Institution, Open Label, Phase II: The protocol was a Single Arm study in which eligible patients were women with a diagnosis of invasive breast cancer with primary or recurrent gross disease in the breast or chest wall or lymph nodes that is progressive, persistent, or minimally responsive to chemotherapy. Patients will received 825 mg/m2 bid of capecitabine. One of the two daily doses of capecitabine will be taken 2 hours before receiving radiotherapy. Capecitabine will be administered when patients receives radiation therapy. Traditional therapy dosage will be 50-57 GY to the initial clinical target volume.
Period: Overall Study
Arm/Group | Single Arm Institution, Open Label, Phase II
Started | 33
Completed | 26
Not Completed | 7
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Insurance Denial | 2

BASELINE CHARACTERISTICS:
Population: Patients who enrolled into the study and signed consent.
Groups:
- Single Arm Institution, Open Label, Phase II: The protocol was a Single Arm study in which eligible patients were women with a diagnosis of invasive breast cancer with primary or recurrent gross disease in the breast or chest wall or lymph nodes that is progressive, persistent, or minimally responsive to chemotherapy. Patients will received 825 mg/m2 bid of capecitabine. One of the two daily doses of capecitabine will be taken 2 hours before receiving radiotherapy. Capecitabine will be administered when patients receives radiation therapy. Tradition therapy does will be 50-57 Gy to the initial clinical target volume.
Arm/Group | Single Arm Institution, Open Label, Phase II
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12.02326)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
  Hungary | 1
  Puerto Rico | 1
  Norway | 1
Patients enrolled were female gender over the age of 18. [Number; unit: participants] — Number of patients enrolled into the protocol were eligible patients who were women over the age of 18.
  participants | 33

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Patients Who Receive Pre-operative or Palliative Concurrent Radiation w/ Capecitabine to the Breast & at Risk or Involved Regional Lymph Nodes Basins.
Description: The response by RECIST was assessed after 45 Gy of radiation for patients with breast cancer treated with concurrent capecitabine and radiation therapy.
Time Frame: Participants were monitored from 2009 to 2012.
Population: All patients who received protocol - specified treatment.
Measure: Number; unit: participants
Groups:
- Single Arm Institution, Open Label, Phase II: Patients will received 825 mg/m2 bid of capecitabine. One of the two daily doses of capecitabine will be taken 2 hours before receiving radiotherapy. Capecitabine will be administered when patients receives radiation therapy. Radiation therapy doses will be 50-57 Gy to the initial clinical target volume.
Arm/Group | Single Arm Institution, Open Label, Phase II
Number analyzed (Participants) | 33
participants | 26

ADVERSE EVENTS:
Time Frame: Subjects will be followed ever 3 months (+/- 1 mo) post-treatment times 1, then every 6 months (+/- 1 mo) times 1, then every 12 months (+/- 2 mos) times 2, up to 3 years
Description: Adverse Events were collected on an excel spreadsheet which captured the start date of the AEs, the description of the AEs and the grade of the AEs.
Arm/Group | Single Arm Institution, Open Label, Phase II
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 18/26
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Institution, Open Label, Phase II (N=26)
Opportunistic Infection (Infections and infestations) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Pulmonary Inflitrates (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 2
Infection with Normal Neutropenia (Blood and lymphatic system disorders) | 3
Edema, limb (Musculoskeletal and connective tissue disorders) | 3
Edema, trunk (Musculoskeletal and connective tissue disorders) | 3
Pain: extremity (Musculoskeletal and connective tissue disorders) | 4
Pain: chest wall (Musculoskeletal and connective tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pain: bone (Musculoskeletal and connective tissue disorders) | 3
Nausea (General disorders) | 4
Pain: esophagus (Gastrointestinal disorders) | 4
Esophagitis (Gastrointestinal disorders) | 4
Pain: lymph node (Blood and lymphatic system disorders) | 4
Pain: skin (Skin and subcutaneous tissue disorders) | 5
Infection with uknown Neutropenia (Blood and lymphatic system disorders) | 5
Thrombus (Blood and lymphatic system disorders) | 6
Vomitting (General disorders) | 7
Pain: stomach (Gastrointestinal disorders) | 7
Hand/foot skin reaction (Skin and subcutaneous tissue disorders) | 6
Diarrhea (Metabolism and nutrition disorders) | 1
Dehydration (Nervous system disorders) | 2
Fatigue (Endocrine disorders) | 1
Fibrosis Deep Connective Tissue (Blood and lymphatic system disorders) | 1
Pain - Cardiac (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT00916578/Prot_SAP_000.pdf